CLINICAL TRIAL: NCT05214183
Title: Acalabrutinib and Rituximab in Elderly Patients With Untreated Mantle Cell Lymphoma
Acronym: ALTAMIRA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic Lymphoma Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG-MCL8 ALTAMIRA
Record Dates: First submitted 2021-10-20; First posted 2022-01-28 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: MCL; Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib-rituximab in patients with untreated mantle cell lymphoma (Experimental)
  Interventions: Drug: Acalabrutinib-rituximab in patients with untreated mantle cell lymphoma

INTERVENTIONS:
Drug: Acalabrutinib-rituximab in patients with untreated mantle cell lymphoma — Acalabrutinib, or ACP-196, is a next generation BTK inhibitor, more selective than ibrutinib, and without in vitro antagonism of anti-CD20 directed immunotherapies, indicating that its combination with rituximab may be more active than the combination of ibrutinib and rituximab

SUMMARY:
This is a phase II trial, with the aim of developing a chemotherapy-free regimen for untreated patients with mantle cell lymphoma (MCL).

Acalabrutinib (ACP-196) is a next generation bruton tyrosine kinase (BTK) inhibitor, more selective than ibrutinib, and without in vitro antagonism of anti-CD20 directed immunotherapies, indicating that its combination with rituximab may be more active than the combination of ibrutinib and rituximab.

In this trial proposal, we will also assess the activity of this combination in comparison to a historical control of ibrutinib + rituximab, consisting of the experimental arm of ibrutinib + rituximab in the randomized ENRICH trial (EudraCT number 2015-000832-13), and data from our previous trial with R-bendamustine-lenalidomide (NLG-MCL4).

The duration of treatment will be a minimum of 12 months. Patients in molecular remission in blood and bone marrow and in complete remission according to CT, will then stop acalabrutinib, but continue on rituximab for a maximum of 36 months. Patients that are minimal residual disease positive (MRD+) will be evaluated again every 6 months and continue on acalabrutinib for a maximum of 36 months.

Patients without a molecular marker, that cannot be followed with MRD, will stop treatment if in CR with PET at 12 months, and be followed by PET-CT every 6 months for a maximum of 36 months.

Patients who convert back to MRD positive after stopping acalabrutinib are reinstalled on acalabrutinib until progression.

Patients with TP53 aberrations and/or blastoid histology, will monitor MRD but continue with treatment until progression regardless of MRD results.

A planned interim analysis will be performed when 40 patients have undergone response assessment after 6 months, for futility and efficacy.

If less than 16 of 40 patients obtain a CR, the trial will be stopped due to futility.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥60 years
2. Pathologically confirmed MCL (according to the 2016 WHO classification), with documentation of monoclonal B cells that have a chromosome translocation t(11;14)(q13;q32) and/or overexpress cyclin D1
3. Stage II-IV, measurable by imaging and requiring treatment in the opinion of the treating clinician
4. No previous treatment for MCL (other than localised radiotherapy or 7-day pulse of steroids for symptom control)
5. ECOG performance status 0 - 2
6. Absolute neutrophil count (ANC) > 1.0 x 109 and platelet count >100 x 109, unless related to lymphoma - in this situation, the threshold for inclusion is ANC > 0.5 x 109 and platelet count > 50 x 109
7. Creatinine clearance > 30 ml/min (Cockcroft-Gault)
8. AST and/or ALT <3xULN and/or total bilirubin <3xULN
9. Able to give voluntary written informed consent
10. Woman of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and for 2 days after the last dose of acalabrutinib or for 12 months after last dose of rituximab, whichever is longer

Exclusion Criteria:

1. Patients considered fit enough to undergo autologous or allogeneic stem cell transplant for MCL
2. Major surgery within two weeks prior to day 1 of cycle 1
3. Patients who are unable to swallow capsules, or who have disease significantly affecting gastrointestinal function that would limit oral absorption of medication
4. Known serological positivity for HBV, HCV, HIV. Patients who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR) result. Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Patients who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded
5. Diagnosed with or treated for any other malignancy than MCL within 2 years prior to day 1 of cycle 1 (except basal cell carcinoma, cutaneous squamous cell carcinoma or any other in situ malignancy)
6. Active infection requiring treatment
7. Serious medical or psychiatric illness likely to interfere with participation in this clinical study
8. Concurrent treatment with another investigational agent outside of this protocol
9. Known history of drug-specific hypersensitivity or anaphylaxis to rituximab or acalabrutinib (including active product or excipient components).
10. Active bleeding, history of bleeding diathesis (eg, hemophilia or von Willebrand disease)
11. Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura)
12. The use of strong CYP3A inhibitors within 1 week or strong CYP3A inducers within 3 weeks of the first dose of study drug is prohibited
13. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon) within 7 days of first dose of study drug
14. Prothrombin time/INR or aPTT (in the absence of Lupus anticoagulant) > 2x ULN
15. Requires treatment with proton pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Patients receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study
16. History of significant cerebrovascular disease or event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug
17. Breastfeeding or pregnant women
18. Concurrent participation in another therapeutic clinical trial
19. History of or ongoing confirmed progressive multifocal leukoencephalopathy (PML)
20. Significant cardiovascular disease such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification at Screening. Note: Subjects with controlled, asymptomatic atrial fibrillation are allowed to enroll on study
21. Received a live virus vaccination within 28 days of first dose of study drug

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 5 years
  The primary efficacy endpoint is progression-free survival, compared to the MCL4 data by log rank test

CONTACTS AND LOCATIONS:
Overall Officials: Mats Jerkeman, Principal Investigator — Department of Oncology, Skåne University Hospital
Locations (20):
- Denmark (2):
  - Department of Hematology X, Odense University Hospital, Odense
  - Department of Hematology, Zeeland University Hospital Roskilde, Roskilde
- Finland (2):
  - Department of Hematology, Helsinki University Hospital Comprehensive Cancer Center, Helsinki
  - Oulu University Hospital, Oulu
- Norway (4):
  - Department of Oncology, Haukeland University Hospital, Bergen
  - Avd. for Kreftbehandling, Oslo Universitetssykehus, Oslo
  - Avdeling for Blod- og Kreftsykdommer, Stavanger Universitetssykehus, Stavanger
  - Kreftklinikken, St Olavs Hospital, Trondheim
- Division of Hematology-Oncology Samsung Medical Center Seoul, Seoul, South Korea
- Sweden (11):
  - Hematological Department, Falu Hospital, Falun, Falun
  - Department of Hematology and Coagulation, Sahlgrenska University Hospital, Gothenburg
  - Department of Medicine, Halmstad Country Hospital, Halmstad
  - Department of Internal Medicine, Kalmar County Hospital, Kalmar
  - Hematologiska Kliniken, Universitetssjukhuset, Linköping
  - Department of Medicine, Sunderbyn Hospital, Luleå
  - Mats Jerkeman, Lund
  - Center of Hematology, Karolinska University Hospital, Stockholm
  - Uddevalla Hospital, Uddevalla
  - Cancercentrum, Norrlands Universitetsjukhus, Umeå
  - Department of Oncology, Uppsala Academic Hospital, Uppsala